CLINICAL TRIAL: NCT02573571
Title: Scoring Personalized Needs in Clostridium Difficile Infections for Fidaxomixin Therapy
Brief Title: Personalized Needs in Clostridium Difficile Infections
Acronym: SPECIFY
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Collaborators: Hellenic Sepsis Study Group (Other)
Responsible Party: Principal Investigator, Evangelos J. Giamarellos-Bourboulis, M.D., Associate Professor of Internal Medicine, University of Athens
Other Study IDs: CL01
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Biologic Markers; Clinical Markers
Keywords: single nucleotide polymorphisms; cytokines; microbiome
MeSH Terms: interventions — Polymorphism, Single Nucleotide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for human DNA extraction and human stool for whole bacterial DNA extraction. Sampling is done on the first day and on disease recurrence
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Clostridium difficile infection: Patients with Clostridium difficile-associated diarrhea for development of biomarkers
  Interventions: Other: Development of biomarkers

INTERVENTIONS:
Other: Development of biomarkers — Blood sampling
  Other Names: Single nucleotide polymorphisms; Serum cytokines

SUMMARY:
To develop a score that can predict early from diagnosis of Clostridium difficile infection (CDI) the risk for relapse and of unfavorable outcome. This score can be used in the future to identify patients will benefit from fidaxomicin treatment.

DETAILED DESCRIPTION:
Medical world is nowadays witnessing a sudden increase of the incidence of infections by Clostridium difficile (DCI). This is due in part to the prolongation of survival of patients with major comorbidities like solid tumor malignancies and lymphomas but also to the widespread intake of proton pump inhibitors and of wide-spectrum antimicrobials. It is highly probable that isolates of C.define causing this pandemic are genetically different than isolates of the same species predominating 20 years ago. This hypothesis is developed based on data of the epidemiology of CDI: in old times administration of clindamycin and ampicillin were the main drivers of CDI; recent studies report fluoroquinolones, 2nd and 3rd generation cephalosporins and even vancomycin (i.e. a drug of choice for CDI) to be linked with the development of CDI.

One major hurdle in management of CDI is relapse; the risk of relapse is reported as 15-20% after the first episode; however it is geometrically increased to even 60-80% after the second episode. As a consequence, management of CDI becomes a major health problem.

Fidaxomicin is a novel compound active against species of C.dificille. Results of two recent double-blind, randomized, large scale clinical studies have shown that oral treatment for 10 days with fidaxomicin 200mg bid was non-inferior to oral treatment with vancomycin 125mg q6h. However, the risk of relapse after treatment with vancomycin was close to 25% and with fidaxomicin close to 15%. This difference was statistically significant in both trials outscoring the superiority of fidaxomicin over vancomycin for the management of CDI. Moreover, meta-analysis has shown a significant reduction in mortality by fidaxomicin.

Despite proven superiority, prescription of fidaxomicin is limited to few cases mostly due to high cost. In many countries prescription is restricted to cases of relapsing CDI. Clinical feeling coming both from post-marketing experience as well as from published evidence supports the use of fidaxomicin for cases with risk of death and overt risk of relapse. However, molecular analysis of the C.difficile pathogen cannot be used as a tool for the prediction of relapse since in relapse cases pathogens carry less than 2 single nucleotide variants of the initial isolate. SPECIFY is aiming to develop a score using both clinical and genetic and biomarker data that can efficiently discriminate patients at risk of severe CDI and at risk of relapse of CDI. This score can become in future a tool to discriminate patients at need for treatment with fidaxomicin instead of traditional treatment with metronidazole/vancomycin.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or more than 18 years
2. Both genders
3. Diarrhea defined as at least 3 episodes of unformed stools in the last 24 hours according to the Bristol stool chart
4. Presence of C.difficile in stool. This is defined as any stool sample positive for the presence of glutamate dehydrogenase (GDH) and for the presence of toxin A and/or B.

Exclusion Criteria:

1. No exclusion criteria exist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Clostridium difficile-associated diarrhea
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Definition of prognostic biomarker | 12 months
  Patients with positive score and unfavorable outcome. Unfavorable outcome is defined as at least one of the following: a) number of patients with severe infection at disease onset; b) number of patients who progress into severe infection; c) number of patients with disease recurrence; and d) number of patients who die

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Skoutelis, MD, Principal Investigator — Evangelismos Athens General Hospital; Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Chair — Attikon Hospital; George Chrysos, MD, PhD, Principal Investigator — Tzaneion Piraeus General Hospital; Styliani Symbardi, MD, PhD, Principal Investigator — Thriassio Elefsis General Hospital; Zoi Alexiou, MD, PhD, Principal Investigator — Thriassio Elefsis General Hospital; Kostantinos Syrigos, MD, PhD, Principal Investigator — Sotiria General Hospital; George Daikos, MD, PhD, Principal Investigator — Laikon Athens General Hospital; Panagiotis Gargalianos, MD, PhD, Principal Investigator — G.Gennimatas Athens General Hospital; Malvina Lada, MD, PhD, Principal Investigator — Sismanogleion General Hospital; Charalambos Gogos, MD, PhD, Principal Investigator — University Hospital of Patras; Ilias Athanasiadis, MD, PhD, Principal Investigator — Mitera General Hospital; Symeon Metallidis, MD, PhD, Principal Investigator — AHEPA Thessaloniki University Hospital
Locations (12):
- Greece (12):
  - 5th Department of Internal Medicine, Evangelismos Athens General Hospital, Athens
  - 1st Department of Internal Medicine, "G.Gennimatas" General hospital, Athens
  - 1st Department of Internal Medicine, Laikon General Hospital, Athens
  - 3rd Department of Internal Medicine, Sotiria General Hospital, Athens
  - 4th Department of Internal Medicine, ATTIKON University Hospital, Athens
  - 2nd Department of Internal Medicine, Sismanogleion General Hospital, Athens
  - 1st Department of Internal Medicine, Thriassio General Hospital, Magoula
  - 2nd Department of Internal Medicine, Thriasio General Hospital, Magoula
  - 2nd Department of Oncology, Mitera Hospital, Marousi
  - Department of Internal Medicine, Patras University Hospital, Pátrai
  - Infections Unit Tzaneion General Hospital, Piraeus
  - 1st Department of Internal Medicine, AHEPA University Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao K, Erb-Downward JR, Walk ST, Micic D, Falkowski N, Santhosh K, Mogle JA, Ring C, Young VB, Huffnagle GB, Aronoff DM. The systemic inflammatory response to Clostridium difficile infection. PLoS One. 2014 Mar 18;9(3):e92578. doi: 10.1371/journal.pone.0092578. eCollection 2014. PMID 24643077
- [Derived] Psarrakis C, Tziolos NR, Matzarakis V, Kumar V, Stylianakis E, Sidiropoulou C, Tasouli E, Iliopoulou K, Samarkos M, Metallidis S, Georgiadou S, Akinosoglou K, Bolanou A, Hatziagelaki E, Kostaki A, Panagopoulos P, Toutouzas K, Milionis H, Adamis G, Poulakou G, Lada M, Skoutelis A, Alexiou Z, Symbardi S, Chrysos G, Netea MG, Giamarellos-Bourboulis EJ. A randomized controlled trial of precision bezlotoxumab treatment for Clostridioides difficile infection. Cell Rep Med. 2026 Jan 20;7(1):102533. doi: 10.1016/j.xcrm.2025.102533. Epub 2026 Jan 2. PMID 41483804